CLINICAL TRIAL: NCT04999137
Title: Evaluation of Pharmacokinetics, Safety and Feasibility for Administration of Two Doses of Intravenous Vitamin C Combined With Vitamin B1 for the Management of Adult Patients Admitted With Sepsis to Kiruddu National Referral Hospital
Brief Title: Evaluation of Safety and Dosing of a Vitamin C Bundle for Sepsis Treatment in Africa
Acronym: REVISTA-DOSE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: Infectious Diseases Institute, Uganda (Other); Walimu (Other); University of Copenhagen (Other); University of Liverpool (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-094
Record Dates: First submitted 2021-04-06; First posted 2021-08-10 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Sepsis; Septic Shock; HIV
Keywords: vitamin c; ascorbate; vitamin b1; thiamine; sepsis; septic shock; hiv; malnutrition
MeSH Terms: conditions — Sepsis; Shock, Septic; Acquired Immunodeficiency Syndrome; Malnutrition | interventions — Ascorbic Acid; Thiamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Intravenous vitamin C 1.5g + intravenous vitamin B1 (Experimental): intravenous vitamin C (1.5 grams) every 6 hours for 16 doses in combination with intravenous vitamin B1 (200 mg) every 12 hours
  Interventions: Drug: Vitamin C; Drug: Vitamin B1
- Intravenous Vitamin C 3g + intravenous vitamin B1 (Experimental): Intravenous vitamin C (3 grams) every 6 hours for 16 doses in combination with intravenous vitamin B1 (200 mg) every 12 hours
  Interventions: Drug: Vitamin C; Drug: Vitamin B1
- Usual Care (No Intervention): Usual care

INTERVENTIONS:
Drug: Vitamin C — Vitamin C (ascor), infused intravenously in 50 mls sodium chloride (NaCl) over 30 minutes every 6 hours for 16 doses
  Other Names: Ascor; Ascorbate
  Arms: Intravenous Vitamin C 3g + intravenous vitamin B1; Intravenous vitamin C 1.5g + intravenous vitamin B1
Drug: Vitamin B1 — Vitamin B1 (200 mg) administered intravenously every 12 hours for 8 doses
  Other Names: Thiamine; Thiamin
  Arms: Intravenous Vitamin C 3g + intravenous vitamin B1; Intravenous vitamin C 1.5g + intravenous vitamin B1

SUMMARY:
Open-label phase 2a Randomized Controlled Trial (RCT) assessing the pharmacokinetics of two different doses of intravenous vitamin C given alongside vitamin B1 in adult medical patients with sepsis and hypotension.

DETAILED DESCRIPTION:
Sepsis is a life-threatening infection which, due to a dysregulated host response to infection, is responsible for more than 11 million deaths annually, a large percentage of which occur in sub-Saharan Africa (sSA). Emerging research shows promising benefits in treating sepsis patients with "metabolic resuscitation" using combinations of hydrocortisone, intravenous (IV) ascorbic acid (vitamin C) and IV thiamine (vitamin B1), alone or in combination. Studies are currently underway in the USA, Europe, Asia, and South America to understand whether combinations of these medicines or the medicines individually can improve outcomes for patients with sepsis. Although none of these studies are being conducted in sSA, the medicines comprising these metabolic 'bundles' are inexpensive, readily available and relatively safe to administer. It is critical that similar studies are conducted in sSA to evaluate whether or not these inexpensive medicines (or a combination of them) are efficacious for improved survival among patients with sepsis. If these studies prove that these medicines can improve survival from sepsis, there is a large potential to save many lives. Through the Preparation for Randomised Evaluation of a VItamin C bundle for Sepsis Treatment in Africa (REVISTA-Prep) studies, the investigators intend to conduct preliminary research in Uganda to help define parameters for a future RCT aimed at identifying the optimal vitamin C and vitamin B1 combination for improving survival from sepsis among adults in sSA, where resources are constrained, intensive care units are rare and issues like poverty, malnutrition and HIV are common. The study described in this protocol (i.e., REVISTA-DOSE) aims to establish the optimal vitamin C dosing strategy for the future REVISTA-RCT (assessing the efficacy of variations of a treatment bundle comprising vitamin C/B1 and/or hydrocortisone for reducing mortality among adult patients with sepsis in Africa).

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥18 years old) patients presenting to the emergency department of Kiruddu National Referral Hospital (KNRH) with:

   * suspected infection [(any of): temperature >38 degrees Celsius or <36 degrees Celsius or (in the past seven days) fevers, rigors, night sweats or antibiotic use]; AND
   * systolic blood pressure (SBP) <90 mmHg
2. Evidence of a personally signed and dated informed consent document indicating that the subject (or a legal representative) has been informed of all pertinent aspects of the study.
3. Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

1. Pregnant or known active breast feeding
2. Non-severe, localized, uncomplicated infection (e.g., cellulitis with only local symptoms) which is apparent on clinical examination
3. Severe bleeding or hemorrhagic shock
4. Hypotension likely secondary to a cause other than sepsis or sepsis-induced cardiac insufficiency
5. Detainee or prisoner
6. Admission to a surgical or obstetric/gynecological ward
7. Emergency surgery required
8. Previously recruited to the REVISTA-DOSE study
9. History of end stage renal disease requiring dialysis
10. Current symptomatic renal stones or or a previous diagnosis of primary hyperoxaluria or oxalate nephropathy
11. History of allergic reactions to vitamin C or vitamin B1
12. Use of vitamin C at a dose greater than 1 g (oral or intravenous) within 24 hours of screening
13. Chronic disease/illness that, in the opinion of the site investigator, has a lifespan of less than 30 days unrelated to current sepsis diagnosis (e.g., advanced malignancy or neurodegenerative disease).
14. Previous or current enrolment in a trial in which co-enrolment is not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-29 (Estimated); Study Completion 2021-12-29 (Estimated)

PRIMARY OUTCOMES:
change in Vitamin C plasma concentration during the intervention period | during the intervention (days 1-5)
  Vitamin C plasma concentrations will be measured during the intervention period using high-performance liquid chromatography (HPLC) with ultraviolet (UV) analysis and compared to baseline (pre-intervention) concentrations

SECONDARY OUTCOMES:
Oxalate excretion in urine | during the intervention (hours 0-12 and 72-84)
  Urine oxalate levels will be measured through two separate 12 hour urine collections.
Incidence of acute hemolysis | during the intervention (days 0-5)
  Acute hemolysis is defined as:
  1. hemoglobin drop of at least 2.5 g/dl within 24 hours of a study drug; OR
  2. reticulocyte count >2 times upper limit of normal at clinical site lab; AND
  3. at least two of the following:
  i. haptoglobin < lower limit of normal; ii. indirect (unconjugated) bilirubin >2 times upper limit of normal; iii. lactate dehydrogenase (LDH) >2 times upper limit of normal
Enrolment rates | up to 3 months
  Enrolment rates of patients with sepsis and hypotension
Rates of adherence to protocol | during the intervention
  Rates of adherence to protocol for treatment, clinical measurements and follow up

OTHER OUTCOMES:
Change in lactate level | during the intervention (hours 0, 6 and 24)
  A correlate for hypoperfusion (or shock)
Pro-calcitonin clearance (PCT-c) | during the intervention (hours 0, 24 and 72)
  Increasing procalcitonin levels may be an indicator of increased severity of bacterial infection or sepsis. PCT-c calculated using the following formula: initial PCT minus PCT at 0 and 24 and 72 hours, divided by the initial PCT multiplied by 100.
Duration of hypotension assessed by systolic and mean arterial pressures during 4-day administration of vitamin C (in combination with vitamin B1) | during the intervention (hours 0-96)
  Lower blood pressures are associated with worsening shock and poor organ perfusion. Non invasive blood pressure readings will be recorded.
Change in quick sepsis related organ failure assessment (qSOFA) score | during the intervention (hours 0, 6, 24, 48, 72 and 96)
  qSOFA score is a 3 point measurement of sepsis severity made up of systolic blood pressure under 100 mmHg, Glasgow Coma Scale (GCS) score <15 and respiratory rate >22. Scores increase with severity from 0-3.
Change in Universal Vital Assessment (UVA) score | during the intervention (hours 0, 6, 24, 48, 72 and 96)
  The UVA score includes points for temperature, heart and respiratory rates, systolic blood pressure, oxygen saturation, GCS score and HIV serostatus. Patients are scored from zero to 13 with increasing severity
Change in Modified Early Warning Score (MEWS) | during the intervention (hours 0, 6, 24, 48, 72 and 96)
  MEWS is a physiologic scoring system for bedside assessment of patients. Patients are scored from 0-14 with increasing severity according to systolic blood pressure, heart rate (HR), respiratory rate (RR), temperature and the 'alert, verbal, pain, unresponsive' (AVPU) score
Percentage of patients able to walk independently | before, during and after the intervention (days 0, 1, 2, 3, 4 and 28)
  Walking independently is defined by being able to stand independently and walk at least 10 steps without assistance
Change in creatinine levels | before, during and after the intervention (days 0, 1, 3 and 28)
  measure of kidney function comparing baseline to measurement during and after the intervention
mortality at 28 days | after the intervention (day 28)
  Number of participants alive 28 days after enrolment
in-hospital mortality | after the intervention (day 7 or at the time of hospital discharge)
  Number of participants alive at hospital discharge (or day 7 if still an inpatient)
mortality at 28 days among vitamin B1 deficient participants | after the intervention (day 28)
  Number of vitamin B1 deficient participants alive 28 days after enrolment
in-hospital mortality among vitamin B1 deficient participants | after the intervention (day 7 or at the time of hospital discharge)
  Number of vitamin B1 deficient participants alive at hospital discharge (or day 7 if still an inpatient)
number of oxygen-free days | during the intervention (days 1-5)
  number of days of hospitalization during which the participant does not require supplemental oxygen for hypoxia and/or respiratory distress
length of hospitalization | during the intervention (days 1-5)
  number of days hospitalized
number of hospital-free days | during and after the intervention (days 1-28)
  taken from 28 days; deceased patients will be assigned a score of 0 for all "free day" outcomes
Frequency of re-admission to hospital | after the intervention (day 28)
  Number of re-hospitalizations after discharge from initial hospitalization for sepsis
change in Vitamin C plasma concentration at day 28 | after the intervention (day 28)
  Vitamin C plasma concentrations will be measured after the intervention period (at 28 days post enrolment) using HPLC with UV analysis and compared to baseline (pre-intervention) concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Shevin T Jacob, MD MPH, Principal Investigator — LSTM/IDI/Walimu
Locations (2):
- Uganda (2):
  - Infectious Diseases Institute, Makerere University, Kampala
  - Kiruddu National Referral Hospital, Kampala

REFERENCES:
- See also: Related Info — https://www.lstmed.ac.uk/ARCS
- See also: Related Info — https://walimu.org/
- See also: Related Info — https://idi.mak.ac.ug/